CLINICAL TRIAL: NCT01952015
Title: A Multi-center, Open Label Study of Subcutaneous Secukinumab in Prefilled Syringes as Mono- or Co-therapy to Assess the Efficacy, Safety and Tolerability in Japanese Subjects With Generalized Pustular Psoriasis
Brief Title: Study to Assess the Efficacy, Safety and Tolerability of Secukinumab in Japanese Subjects With Generalized Pustular Psoriasis (GPP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A1302
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Psoriasis
Keywords: generalized pustular psoriasis; skin condition; skin disease,
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AIN457 (Experimental): All subjects were assigned to receive 150 mg secukinumab (AIN457) by subcutaneous injections. AIN457 was administered at baseline, weeks 1, 2, 3, 4. Prior to receiving the week 8 dose, all subjects were assigned to the following treatment group based on clinical components of their Clinical Global Impression (CGI) evaluation at week 8.
  * "No up-titration" group received 1 injection of 150 mg AIN457 at weeks 8, 12, and each visit from week 16 until week 48.
  * "Up-titration" group received 2 injections of 150 mg AIN457 at weeks 8, 9, 12 and each visit from week 16 until week 48.
  Subjects who received 150 mg AIN457 can be up-titrated to 300 mg AIN 457 at any visit starting at week 16 based on clinical components of their CGI evaluation and investigator's discretion.
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — Secukinumab (AIN457) 150 mg, provided in a 1 mL prefilled syringe (one syringe for 150 mg dose, two syringes for the 300 mg dose).

SUMMARY:
The purpose of this study was to assess efficacy and safety data of secukinumab in Japanese subjects with generalized pustular psoriasis (GPP). This study was expected to support the filing of secukinumab in the indication of pustular psoriasis in Japan.

ELIGIBILITY:
Inclusion Criteria:

* At baseline, presence of GPP classified on the basis of the criteria for diagnosis of GPP by Japanese Dermatological Association (JDA)
* At baseline, erythema area with pustule ≥ 10%

Exclusion Criteria:

* Erythrodermic, guttate psoriasis, or subcorneal pustular dermatosis at screening.
* At baseline, : total score of JDA severity index for GPP ≥ 14
* Drug-induced psoriasis
* Ongoing use of prohibited psoriasis treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08-21 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Inashiki-gun, Ibaraki
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 patients were screened, and 12 patients entered the induction period. The reason for all screen failures was patient/guardian decisions
Period: Induction
Arm/Group | AIN457
Started | 12
Completed | 11
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Maintenance
Arm/Group | AIN457
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 2
Period: Treatment Period 3
Arm/Group | AIN457
Started | 9
Completed | 0
Not Completed | 9
Not completed — Physician Decision | 9

BASELINE CHARACTERISTICS:
Population: Safety set: The safety set included all patients who took at least one dose of study treatment during the treatment period.
Arm/Group | AIN457
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (15.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Success at Week 16 Using Non-responder Imputation (Full Analysis Set)
Description: Treatment success was defined as "Minimally improved", "Much improved" or "Very much improved" in Clinical global impression (CGI).
  Non-responder imputation assigns a value of nonresponse to missing data points, any patient who drops out is assumed to be a non-responder.
Time Frame: 16 weeks
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Number; unit: Participants
Arm/Group | AIN457
Number analyzed (Participants) | 12
Participants
  Treatment success - Yes | 10
  Treatment success - No | 2
  Very much improved | 9
  Much improved | 1
  Minimally improved | 0
  No change | 1
  Worse | 0
  Missing | 1

2. Secondary Outcome: Number of Patients With Treatment Success at Week 52 Using Non-responder Imputation (Full Analysis Set)
Description: Ten patients showed treatment success at week 52 with clinical global impression (CGI) evaluated as "very much improved", "much improved", "minimally improved".
  Two patients did not achieve treatment success at week 52 with CGI evaluated as "missing" and both were imputed as "no treatment success".
Time Frame: 52 weeks
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Number; unit: Participants
Arm/Group | AIN457
Number analyzed (Participants) | 12
Participants
  Treatment success - Yes | 10
  Treatment success - No | 2
  CGI - very much improved | 7
  CGI - much improved | 2
  CGI - minimally improved | 1
  CGI - No change | 0
  CGI - worse | 2

3. Secondary Outcome: Number of Patients With Treatment Success at End of Trial Using Non-responder Imputation (Full Analysis Set)
Description: Clinical global impression (CGI) evaluated as "very much improved", "much improved", "Minimally improved".
Time Frame: week 148
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Number; unit: Participants
Arm/Group | AIN457
Number analyzed (Participants) | 12
Participants
  Very much improved: number analyzed (Participants) | 9
  Very much improved | 8
  Much improved: number analyzed (Participants) | 9
  Much improved | 1
  Minimally improved: number analyzed (Participants) | 9
  Minimally improved | 0
  No change: number analyzed (Participants) | 9
  No change | 0
  Worse: number analyzed (Participants) | 9
  Worse | 0
  Missing: number analyzed (Participants) | 9
  Missing | 0

4. Secondary Outcome: Summary of Clinical Global Impression up to End of Trial
Description: Clinical Global Impression (CGI) has five categories: Very much improved, much improved, minimally improved, no change and worsened.
  Two patients did not achieve treatment success at week 52 with CGI evaluated as missing and both were imputed as "no treatment success".
Time Frame: up to week 148 (End of Trial)
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Number; unit: Participants
Groups:
- Very Much Improved; Much Improved; Minimally Improved; No Change; Worse; Missing: All subjects were assigned to receive 150 mg secukinumab (AIN457) by subcutaneous injections.
  Clinical global impression (CGI) was evaluated as very much improved, much improved, minimally improved, no change, worse, and missing.
Arm/Group | Very Much Improved | Much Improved | Minimally Improved | No Change | Worse | Missing
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Participants
  Week 1: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
  Week 1 | 4 | 5 | 1 | 1 | 0 | 0
  Week 2: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
  Week 2 | 7 | 4 | 0 | 0 | 0 | 0
  Week 3: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
  Week 3 | 10 | 1 | 0 | 0 | 0 | 0
  Week 4 | 10 | 2 | 0 | 0 | 0 | 0
  Week 8 | 9 | 2 | 0 | 1 | 0 | 0
  Week 16: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
  Week 16 | 9 | 1 | 0 | 1 | 0 | 0
  Week 24: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
  Week 24 | 8 | 1 | 1 | 0 | 1 | 0
  Week 36: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
  Week 36 | 7 | 3 | 0 | 1 | 0 | 0
  Week 52: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
  Week 52 | 7 | 2 | 1 | 0 | 0 | 0
  Week 64: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
  Week 64 | 8 | 1 | 0 | 0 | 0 | 0
  Week 80: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
  Week 80 | 7 | 2 | 0 | 0 | 0 | 0
  Week 96: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
  Week 96 | 8 | 1 | 0 | 0 | 0 | 0
  Week 112: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
  Week 112 | 4 | 1 | 0 | 0 | 0 | 0
  Week 128: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
  Week 128 | 2 | 0 | 0 | 0 | 0 | 0
  Week 140: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
  Week 140 | 8 | 1 | 0 | 0 | 0 | 0

5. Secondary Outcome: Summary of JDA Total Score Category for GPP by Visit up to End of Trial
Description: Japanese dermatological association (JDA) severity index for generalized pustular psoriasis (GPP) included 3 categories (mild, moderate, and severe) in the severity index.
Time Frame: up to week 148 (End of Trial)
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Number; unit: Participants
Groups:
- None; Mild; Moderate; Severe; Missing: All subjects were assigned to receive 150 mg secukinumab (AIN457) by subcutaneous injections. The category of JDA severity index was defined by 3 categories: mild, moderate, and severe.
Arm/Group | None | Mild | Moderate | Severe | Missing
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants
  Baseline | 0 | 9 | 3 | 0 | 0
  Week 1: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
  Week 1 | 0 | 10 | 1 | 0 | 0
  Week 2: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
  Week 2 | 0 | 11 | 0 | 0 | 0
  Week 3: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
  Week 3 | 0 | 11 | 0 | 0 | 0
  Week 4 | 1 | 11 | 0 | 0 | 0
  Week 8 | 0 | 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
  Week 16 | 0 | 11 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
  Week 24 | 1 | 9 | 1 | 0 | 0
  Week 36: number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
  Week 36 | 1 | 10 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Week 52 | 1 | 9 | 0 | 0 | 0
  Week 64: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
  Week 64 | 1 | 8 | 0 | 0 | 0
  Week 80: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
  Week 80 | 3 | 6 | 0 | 0 | 0
  Week 96: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
  Week 96 | 2 | 7 | 0 | 0 | 0
  Week 112: number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
  Week 112 | 0 | 5 | 0 | 0 | 0
  Week 128: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2
  Week 128 | 0 | 2 | 0 | 0 | 0
  Week 144: number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
  Week 144 | 2 | 7 | 0 | 0 | 0

6. Secondary Outcome: The Japanese Dermatological Association (JDA) Component Score for GPP Over Time
Description: The following components of the JDA severity index for generalized pustular psoriasis (GPP) were reported: body surface area (SA)covered with total erythema with pustules, body SA covered with total erythema, body SA covered with edema, fever, white blood cell (WBC) count, C-reactive protein, serum albumin.
  The total score of JDA severity index was assigned a score of 0-17. Assessment of skin lesions: area of erythema with pustules, area of erythema, and area of edema; each score 0-3. Assessment of systemic manifestations and laboratory findings: fever, WBC count, CRP and serum albumin; each score 0-2.
  The higher the JDA severity index for GPP score the worse the outcome.
Time Frame: up to week 148 (end of trial)
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Mean (Standard Deviation); unit: mean scores on a scale
Arm/Group | AIN457
Number analyzed (Participants) | 12
mean scores on a scale
  Body SA w/ erythema with pustules - Baseline | 2 (0.00)
  Body SA w/ erythema with pustules - Week 24: number analyzed (Participants) | 11
  Body SA w/ erythema with pustules - Week 24 | 0.3 (0.65)
  Body SA w/ erythema with pustules - Week 52: number analyzed (Participants) | 10
  Body SA w/ erythema with pustules - Week 52 | 0.0 (0.00)
  Body SA w/ erythema w/ pustules - End of Treatment: number analyzed (Participants) | 9
  Body SA w/ erythema w/ pustules - End of Treatment | 0.0 (0.00)
  Body SA w/ total erythema - Baseline | 1.6 (0.67)
  Body SA w/ total erythema - Week 24: number analyzed (Participants) | 11
  Body SA w/ total erythema - Week 24 | 1.1 (0.54)
  Body SA w/ total erythema - Week 52: number analyzed (Participants) | 10
  Body SA w/ total erythema - Week 52 | 0.8 (0.42)
  Body SA w/ total erythema - End of Treatment: number analyzed (Participants) | 9
  Body SA w/ total erythema - End of Treatment | 0.7 (0.50)
  Body SA w/ edema - Baseline | 1.3 (0.89)
  Body SA w/ edema - Week 24: number analyzed (Participants) | 11
  Body SA w/ edema - Week 24 | 0.4 (0.67)
  Body SA w/ edema - Week 52: number analyzed (Participants) | 10
  Body SA w/ edema - Week 52 | 0.3 (0.48)
  Body SA w/ edema - End of Treatment: number analyzed (Participants) | 9
  Body SA w/ edema - End of Treatment | 0.1 (0.33)
  Fever - Baseline | 0.2 (0.39)
  Fever - Week 24: number analyzed (Participants) | 11
  Fever - Week 24 | 0.2 (0.40)
  Fever - Week 52: number analyzed (Participants) | 10
  Fever - Week 52 | 0.4 (0.52)
  Fever - End of Treatment: number analyzed (Participants) | 9
  Fever - End of Treatment | 0.1 (0.33)
  White blood cell (WBC) count - Baseline | 0.3 (0.65)
  White blood cell (WBC) count - Week 24: number analyzed (Participants) | 11
  White blood cell (WBC) count - Week 24 | 0.1 (0.30)
  White blood cell (WBC) count - Week 52: number analyzed (Participants) | 10
  White blood cell (WBC) count - Week 52 | 0.1 (0.32)
  White blood cell (WBC) count - End of Treatment: number analyzed (Participants) | 9
  White blood cell (WBC) count - End of Treatment | 0.0 (0.00)
  C-reactive protein - Baseline | 0.5 (0.67)
  C-reactive protein - Week 24: number analyzed (Participants) | 11
  C-reactive protein - Week 24 | 0.2 (0.40)
  C-reactive protein - Week 52: number analyzed (Participants) | 10.0
  C-reactive protein - Week 52 | 0.2 (0.42)
  C-reactive protein - End of Treatment: number analyzed (Participants) | 9
  C-reactive protein - End of Treatment | 0.3 (0.50)
  Serum albumin - Baseline | 0.0 (0.00)
  Serum albumin - Week 24: number analyzed (Participants) | 11
  Serum albumin - Week 24 | 0.0 (0.00)
  Serum albumin - Week 52: number analyzed (Participants) | 10
  Serum albumin - Week 52 | 0.1 (0.32)
  Serum albumin - End of Treatment: number analyzed (Participants) | 9
  Serum albumin - End of Treatment | 0.0 (0.00)

7. Secondary Outcome: Change From Baseline in Observed Value of Components of the JDA Severity Index for GPP
Description: The observed value for the following components of the JDA severity index for GPP were reported: percentage of body surface area covered with erythema with pustules, percentage of body surface area covered with total erythema, percentage of body surface area covered with edema, fever (body temperature,°C), white blood cell (WBC) count (/μL), C-reactive protein (mg/L), serum albumin (g/dL).
  Percent change=100 x Absolute change/post baseline.
Time Frame: up to week 148 (end of trial)
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- AIN457: All subjects were assigned to receive 150 mg secukinumab (AIN457) by subcutaneous injections.
Arm/Group | AIN457
Number analyzed (Participants) | 12
Percent change
  Area of erythema with pustules (Week 24) | -89.09 (33.001)
  Area of erythema with pustules (Week 52) | -100.00 (0.000)
  Area of erythema with pustules (Week 148) | -100.00 (0.000)
  Area of Erythema (Week 24) | -63.56 (46.693)
  Area of Erythema (Week 52) | -83.60 (24.442)
  Area of Erythema (Week 148) | -87.01 (15.826)
  Area of Edema (Week 24) | -47.92 (107.200)
  Area of Edema (Week 52) | -69.17 (69.733)
  Area of Edema (Week 148) | -99.05 (2.520)
  Body temperature (Week 24) | -0.27 (1.071)
  Body temperature (Week 52) | 0.08 (1.076)
  Body temperature (Week 148) | -0.87 (1.473)
  WBC (Week 24) | -15.16 (23.120)
  WBC (Week 52) | -22.16 (28.009)
  WBC (Week 148) | -25.63 (18.838)
  CRP (Week 24) | 18.12 (197.270)
  CRP (Week 52) | 34.21 (245.564)
  CRP (Week 148) | 30.60 (146.990)
  Serum Albumin (Week 24) | 0.73 (7.952)
  Serum Albumin (Week 52) | 0.63 (12.952)
  Serum Albumin (Week 148) | 1.64 (3.688)

8. Secondary Outcome: Mean Health-related Quality of Life (The Dermatology Life Quality Index [DLQI] and Short Form Health Survey [SF-36]) Over Time
Description: DLQI is a 10-item general dermatology disability index designed to assess HRQL in adults with skin diseases (Finlay & Khan 94). The measure is self-admin. & includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. DLQI total score is the sum of the 10 questions. Each item has four response categories, ranging from 0 (not at all) to 3 (very much). Scores range from 0 to 30 9higher scores indicate greater health-related quality of-life impairment). SF-36 is a widely used and extensively studied instrument to measure HRQL among healthy subjects with acute & chronic conditions (Ware et al. 93, 94). It consists of 8 subscales (based on a scale of 0-100) that can be scored individually: Two overall summary scores for SF-36, the Physical Component Summary (PCS) and the Mental Component Summary (MCS), were computed. DLQI total score decreases and SF-36 increases with improvement of quality of life.
Time Frame: Up to week 148 (end of treatment)
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457
Number analyzed (Participants) | 12
scores on a scale
  DLQI total score at Baseline | 8.4 (6.88)
  DLQI total score at Week 24: number analyzed (Participants) | 11
  DLQI total score at Week 24 | 4.5 (5.16)
  DLQI total score at Week 52: number analyzed (Participants) | 10
  DLQI total score at Week 52 | 2.7 (2.41)
  DLQI total score at end of treatment: number analyzed (Participants) | 9
  DLQI total score at end of treatment | 4.7 (8.25)
  SF-36 - MCS at Baseline | 43.69 (17.472)
  SF-36 - MCS at Week 24: number analyzed (Participants) | 11
  SF-36 - MCS at Week 24 | 46.70 (9.9696)
  SF-36 - MCS at Week 52: number analyzed (Participants) | 10
  SF-36 - MCS at Week 52 | 46.27 (11.768)
  SF-36 - MCS at end of trial: number analyzed (Participants) | 9
  SF-36 - MCS at end of trial | 47.70 (13.457)
  SF-36 - PCS at Baseline | 50.61 (3.258)
  SF-36 - PCS at Week 24: number analyzed (Participants) | 11
  SF-36 - PCS at Week 24 | 52.39 (4.438)
  SF-36 - PCS at Week 52: number analyzed (Participants) | 10
  SF-36 - PCS at Week 52 | 50.20 (4.670)
  SF-36 - PCS at end of treatment: number analyzed (Participants) | 9
  SF-36 - PCS at end of treatment | 49.82 (6.528)

9. Secondary Outcome: Number of Patients With GPP-related Systemic and Topical Co-medication Over Time
Description: Use of systemic and topical co-medication to treat generalized pustular psoriasis (GPP), in subjects who have active GPP treatment at baseline.
Time Frame: up to week 52
Population: Full analysis set (FAS): The FAS was comprised of all patients who entered into the induction period.
Measure: Number; unit: Participants
Arm/Group | AIN457
Number analyzed (Participants) | 12
Participants
  Topical co-medication related to GPP | 12
  Systemic co-medication related to GPP | 8

ADVERSE EVENTS:
Time Frame: Adverse events are collected from first patient first visit (FPFV) until last patient last visit (LPLV). All adverse events reported in this record are from the late of first patient first treatment until last patient last visit, approximately 3 years.
Description: AE additional description
Arm/Group | AIN457
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 (N=12)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
CELLULITIS (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 1
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1
CATARACT (Eye disorders) | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
DUODENITIS (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1
PYREXIA (General disorders) | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
CELLULITIS (Infections and infestations) | 1
ECZEMA IMPETIGINOUS (Infections and infestations) | 1
ERYTHRASMA (Infections and infestations) | 1
FOLLICULITIS (Infections and infestations) | 1
GENITAL CANDIDIASIS (Infections and infestations) | 1
HELICOBACTER INFECTION (Infections and infestations) | 1
IMPETIGO (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 7
OTITIS EXTERNA (Infections and infestations) | 1
PARONYCHIA (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
STREPTOCOCCAL INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BURNING SENSATION (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1
SOMNOLENCE (Nervous system disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
BREAST CYST (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 1
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 1
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 1
PURPURA SENILE (Skin and subcutaneous tissue disorders) | 1
SOLAR DERMATITIS (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigators from publishing. Any publications from a single-site are postponed until the publication of the pooled data (o.e., data from all sites) in the clinical trial.